CLINICAL TRIAL: NCT00147628
Title: A Multi-Center, Double-Blind Placebo Controlled, Flexible-Dose Study With An Open-Label Phase To Assess The Efficacy Of Sildenafil Citrate On Erectile Function And Intercourse Satisfaction As Well As To Validate The Sexual Experience Questionnaire And Its Treatment Responsiveness In Men With Erectile Dysfunction
Brief Title: Assessment Of Sildenafil On Erectile Function And Intercourse Satisfaction And To Validate A New Subject Questionnaire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481236
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: sildenafil citrate
Drug: placebo for sildenafil citrate

SUMMARY:
To evaluate the effectiveness of sildenafil on erectile function and intercourse satisfaction in men with ED as well as to validate the new Sexual Experience Questionnaire which incorporates functional and emotional elements of a man's sexual experience into one comprehensive questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of erectile dysfunction, defined by a score of less than or equal to 25 on the Erectile Dysfunction domain of the International Index of Erectile Function

Exclusion Criteria:

* Subjects who have been treated with more than 6 doses of sildenafil or any other phosphodiesterase type 5 inhibitor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2005-11; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are: The changes from baseline to Visit 5 (Week 10) of the Erectile Function (Questions 1-5, 15) Intercourse Satisfaction domains (Questions 6-8) of the International Index of Erectile Function (IIEF).

SECONDARY OUTCOMES:
The change from baseline to Visit 4 (Week 6), Visit 5 (Week 10) and Visit 7 (Week 16) in the domains and total score as well as the individual questions of the Sexual Experience Questionnaire (SEX-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- [Derived] Kaminetsky JC, Stecher V, Tseng LJ. Quality of erections by age group in men with erectile dysfunction. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.12976. Epub 2017 Sep 11. PMID 28892218
- [Derived] Cappelleri JC, Bushmakin AG, Symonds T, Schnetzler G. Scoring correspondence in outcomes related to erectile dysfunction treatment on a 4-point scale (SCORE-4). J Sex Med. 2009 Mar;6(3):809-19. doi: 10.1111/j.1743-6109.2008.01155.x. Epub 2009 Jan 7. PMID 19143915
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481236&StudyName=Assessment+Of+Sildenafil+On+Erectile+Function+And+Intercourse+Satisfaction+And+To+Validate+A+New+Subject+Questionnaire